CLINICAL TRIAL: NCT02760511
Title: Anthocyanin Dose-escalation Study in Healthy Young Adults: A CONSORT-compliant, Randomized, Controlled Trial
Brief Title: Anthocyanin Dose-escalation Study in Healthy Young Adults
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaoguan University (Other)
Collaborators: Sun Yat-sen University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: SGU-04
Record Dates: First submitted 2016-04-13; First posted 2016-05-03 (Estimated); Last update posted 2019-03-25 (Actual); Status verified 2016-04

CONDITIONS: Healthy
Keywords: Randomized Controlled Trial; Anthocyanin; Antioxidants
MeSH Terms: interventions — Anthocyanins

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (6):
- Control (Placebo Comparator): Intake of placebo capsules
  Interventions: Dietary Supplement: Placebo
- 20 mg (Active Comparator): Daily intake of 20 mg anthocyanin
  Interventions: Dietary Supplement: Anthocyanin
- 40 mg (Active Comparator): Daily intake of 40 mg anthocyanin
  Interventions: Dietary Supplement: Anthocyanin
- 80 mg (Active Comparator): Daily intake of 80 mg anthocyanin
  Interventions: Dietary Supplement: Anthocyanin
- 160 mg (Active Comparator): Daily intake of 160 mg anthocyanin
  Interventions: Dietary Supplement: Anthocyanin
- 320 mg (Active Comparator): Daily intake of 320 mg anthocyanin
  Interventions: Dietary Supplement: Anthocyanin

INTERVENTIONS:
Dietary Supplement: Anthocyanin — Capsules with different anthocyanin content
  Arms: 160 mg; 20 mg; 320 mg; 40 mg; 80 mg
Dietary Supplement: Placebo — Placebo capsules
  Arms: Control

SUMMARY:
Anthocyanins are naturally existing, polyphenolic compounds found in the vacuolar sap of the epidermal tissues of flowers and fruits, with a pink, red, blue, or purple color. Recently, study of anthocyanin pigments has drawn more and more interest since several epidemiological studies have demonstrated their health-promoting properties, such as reducing lipid accumulation and decreasing oxidative stress and inflammation. Nevertheless, there is a clear need for advancing understanding with regard to effective amounts of intake for these phytochemicals. The aim of this study was to investigate the efficacy and pharmacokinetics of anthocyanin in healthy volunteers.

ELIGIBILITY:
Inclusion Criteria:

* Blood test, liver function test, renal function test are normal;
* Blood lipids, cardiac function are normal;
* 18.5<BMI<23.9;
* Regular dietary, seldomly eating outside;
* Stable condition of body weight in recent 3 months

Exclusion Criteria:

* > 140 grams of alcohol/week for male and >70 grams of alcohol/week for female, smoking regularly;
* Known diagnosis of acute diseases or chronic diseases in recent 1 month;
* Be planning to be pregnant in a year, or being pregnant and lactation.

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 122 (Actual)
Dates: Start 2016-02-01 (Actual); Primary Completion 2016-09-01 (Actual); Study Completion 2017-05-01 (Actual)

PRIMARY OUTCOMES:
Plasma total antioxidant capacity | 2 weeks
  Oxidative stress
Plasma malondialdehyde concentrations | 2 weeks
  Oxidative stress
Plasma 8-iso-prostaglandin concentrations | 2 weeks
  Oxidative stress

SECONDARY OUTCOMES:
Plasma tumor necrosis factor alpha concentrations | 2 weeks
  Inflammatory response
Plasma interleukin-6 concentrations | 2 weeks
  Inflammatory response

CONTACTS AND LOCATIONS:
Locations (1):
- Shaoguan University, Shaoguan, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided